CLINICAL TRIAL: NCT05491174
Title: Feasibility and Acceptability of a Randomised Controlled Trial, Examining a Transdiagnostic DBT-informed Skills Group Intervention Delivered by Protocolised Based Intervention Facilitators (P-BIFS) for Adults in Community Mental Health Settings
Brief Title: Mental Health Intervention for Transdiagnostic Groups in the Community
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King's College London (Other)
Collaborators: South London and Maudsley NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: R&D2022/045
Record Dates: First submitted 2022-07-29; First posted 2022-08-08 (Actual); Last update posted 2023-10-03 (Actual); Status verified 2023-09

CONDITIONS: Severe Mental Illness
Keywords: Severe Mental Illness; Dialectical Behavioural Therapy; Emotion Regulation
MeSH Terms: conditions — Mental Disorders; Emotional Regulation

STUDY DESIGN:
Intervention Model Description: Participants are assigned to either the intervention arm (DBT-informed skills group) or a wait-list control.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DBT-Informed Intervention (Experimental): The DBT-informed group intervention, known as the 'Managing Emotions Group', will consist of 90-minute sessions, run weekly over 10 weeks.
  Interventions: Behavioral: DBT-Informed skills group
- Wait-list control (No Intervention): Participants will be placed on a wait-list for up to 18 weeks.

INTERVENTIONS:
Behavioral: DBT-Informed skills group — 10 session group ran weekly by junior staff (P-BIFs) following a standardised manual-based protocol which can be delivered either face-to-face or via video-call. The groups will be skills-based, covering each of the four modules of DBT: Mindfulness, Distress Tolerance, Emotion Regulation and Interpersonal Effectiveness.
  Other Names: Managing Emotions Group
  Arms: DBT-Informed Intervention

SUMMARY:
The investigators propose to evaluate a new protocol-based intervention that is informed by Dialectical Behaviour Therapy (DBT), known as a DBT-informed intervention, delivered in routine mental health settings within South London and Maudsley NHS foundation trust. The intervention is delivered to a group of transdiagnostic service users with a severe mental illness (SMI). It is delivered by a junior workforce who will be referred to as Protocol-Based Intervention Facilitators (P-BIFs). Successful delivery by a less expert workforce has potential to increase routine implementation, compared to delivery by expert staff, where costs of both salary and training are higher.

Dialectical Behaviour Therapy (DBT) is a type of psychological treatment recommended for people with a diagnosis of emotionally unstable personality disorder (EUPD). Individuals with a diagnosis of EUPD commonly experience difficulties with managing and responding to their emotions. This is known as emotion dysregulation. Difficulties with emotion dysregulation are thought to play a role in many mental health difficulties. The evidence base for using interventions that are informed by DBT, known of as DBT informed interventions with other mental health diagnoses, is emerging.

The current research aims to investigate whether it is possible (feasible) to conduct a randomised control trial evaluating the transdiagnostic DBT-informed skills group for individuals representative of SMI presentations seen within community mental health settings. The study will also examine whether it is possible for junior staff to deliver the manualised group intervention.

Service user participants will be randomised to either a 10-week DBT-informed intervention delivered by the P-BIFs, or a waitlist. Those on the waitlist will access the intervention once their involvement in the study has ended. The study will last for up to 1 year. The maximum duration to complete trial participation from consent to completion will be 18 weeks.

It is hypothesized that the DBT informed intervention, delivered by junior staff, will be feasible and acceptable with this client population.

DETAILED DESCRIPTION:
Primary objectives of the research are:

1. To determine the feasibility and acceptability of conducting a double-arm randomised control trial (RCT) of a transdiagnostic Dialectical Behavioural Therapy informed (DBT-informed) group intervention within secondary care mental health settings.
2. To determine feasibility and acceptability of training Protocol Based Intervention facilitators (P-BIFs), to deliver the intervention as per the protocol.

   Feasibility will be measured using pre-specified criteria.

   A secondary objective is to explore change in assessment scores between the treatment and control group.

   The research will utilise an experimental, open-label double-arm randomised design investigating feasibility. Service user participants will be randomly allocated to either the intervention group or the waitlist control group using randomisation software. Pairwise randomisation will be used whereby participants will be randomised in pairs for an approximately equal number of participants in each arm.

   Baseline measures (T0) are completed by all service-user participants before randomisation occurs to ensure both participants and researchers are blinded. Once randomised, participants will be unblinded but subsequent measures will be completed with a staff member unaware of allocation to minimise bias. The questionnaire pack is completed again by all participants at 18 weeks (T18, end of intervention and waitlist). Feasibility will be assessed by predetermined count data and P-BIF adherence to the protocolised intervention.

   Recruitment: Both service user and P-BIF participants will be recruited from recovery services with South London and Maudsley (SLaM) NHS Foundation Trust, specifically Lambeth Adult Mental Health services

   Trial participation procedure:

   Service users: After receiving informed consent, the researcher will access medical records in order to collect demographic information.

   Participants will then be asked to complete the baseline assessment questionnaire pack either independently, or with a member of the clinical team (who is not involved in the delivery of the group the participant will attend) if requested.

   The research team will examine the completed questionnaire pack for any missed questions or errors (e.g. selecting more than one response to a question that only requires a single response). Where this is the case, the researcher will arrange a telephone call with the participant to confirm their responses ensuring full data sets are obtained.

   The participant will then be randomised into one of two groups. Group A will receive the group intervention and Group B will act as a waitlist control group.

   Participants randomised to the treatment arm (Group A):

   Participants randomised to the treatment arm will commence treatment in the next available treatment group.

   Participants in Group A will be expected to attend weekly, 90-minute sessions for 10 weeks. Once the 10-week intervention is complete, participants in the treatment arm will be asked to complete the assessment pack (T18). Once T18 assessment measures are completed, their involvement in the study will end.

   Participants randomised to waitlist control arm (Group B):

   Participants randomised to the waitlist control will commence their wait period after randomisation. Participants will remain on the treatment waiting list but will not commence the DBT-informed skills group for up to 18 weeks. All other aspects of care will continue as normal. After an 18 week wait, participants in Group B will complete the T18 assessment pack. Once T18 assessment measures are completed, involvement in the study will end. Participants will be offered the intervention as part of usual routine care.

   P-BIFs:

   After informed consent has been received the P-BIFs will be informed about the arrangements for co-facilitating a group by a member of the clinical team.

   P-BIFs will deliver 10, 90-minute weekly sessions following the content and structure outlined in the treatment manual, which includes opportunity for group discussion. After each session, P-BIFs will complete a self-assessment checklist to measure adherence to the protocol.

   Analysis:

   Sample size: The target sample size for service user participants is 30, equating to 15 participants per arm. This is considered sufficient to estimate parameters such as standard deviation for use in sample size calculation in full-scale RCT, whilst accounting for 20% attrition.

   The target sample size for P-BIF participants is between 5 and 10.

   Descriptive analysis: Descriptive statistics will be analysed to ascertain feasibility. Feasibility outcomes will be presented descriptively using measures of central tendency. All participant flow in the study will be reported in accordance with the Consolidated Standards of Reporting Trials (CONSORT) principles.

   Feasibility:

   Predetermined count data:
   1. Recruitment to the target sample of 30 participants (15 per arm), allowing for 20% attrition, so a final target sample of 24 (12 per arm).
   2. Retention rates:

   i. Progression criteria for retention rates will be evaluated using a 'traffic light system'. Retention rates are considered between T0 and T18.

   c. Outcome measure completion rate: i. Progression criteria will also be used for completion of outcome measures. d. Adherence to group intervention: i. Progression criteria will also be used for treatment completion. Completion of the group intervention is operationalised as attending 50% or more of the groups.

   e. Examination of scores on the Satisfaction Questionnaire. 'Neutral' ratings and positive ratings of 'agree' and 'strongly agree' will indicate acceptability of the intervention.

   f. Recruitment to the target sample of between 5 and 10 P-BIFS g. P-BIFs adherence to intervention protocol i. delivery of the intervention must demonstrate adherence to the intervention protocol, as self-rated by the P-BIFs after each session using a checklist. Adherent delivery is defined as meeting ≥90% of checklist.

   ii. P-BIF attendance at supervision will be recorded as an additional measure of treatment adherence.

   Exploration of changes in assessment scores between groups:

   Separate paired t-tests, or Wilcoxon Signed-rank tests (where the assumption of normality has been violated) will be calculated for each outcome measure to explore between-group mean differences. Violations of normality assumptions will be assessed using Shapiro-Wilks test and visual inspection of the relevant histograms and boxplots.

   Due to the exploratory nature of the study, multiple comparisons will not be controlled for. Effect sizes will be reported using Cohen's d (Cohen, 1992) and Pearson r correlation (Cohen, 1988, 1992) with 95% confidence intervals.

   Participant Adherence & Fidelity:

   Participants will need to attend at least one group session to be considered to have attended the intervention. To be considered as having completed the intervention, participants need to attend ≥50% of sessions (considered to reflect a therapeutic dose).

ELIGIBILITY:
Inclusion Criteria for service users:

1. Currently accessing secondary care mental health services within South London and Maudsley NHS Foundation Trust Services, specifically Lambeth Adult Mental Health services.
2. Primary diagnosis considered a severe mental illness according to clinical team.
3. Sufficient English language ability to understand group intervention
4. Anticipate availability for the duration of the study.
5. Capacity to provide informed consent according to clinical team

Inclusion Criteria for P-BIFs:

1. Working at South London and Maudsley NHS Foundation Trust with permission granted by their clinical supervisor to participate.
2. Hold an undergraduate degree in psychology and/or a minimum of 1-year experience working in mental health settings.
3. Capacity to provide informed consent.
4. Have completed, or will complete training to deliver the DBT-informed group intervention as part of routine clinical practice.

Exclusion Criteria for service users:

1. Inability to interact in a group setting for 90 minutes
2. Not available for study duration
3. Difficulties thought to be the result of an organic disorder
4. Lack capacity to consent to participation in the study (assessed by clinical team)
5. Insufficient English language to understand the group intervention

Exclusion Criteria for P-BIFs:

a) Inability to commit for the duration of the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2023-01-27 (Actual); Study Completion 2023-07-20 (Actual)

PRIMARY OUTCOMES:
Feasibility - Recruitment to the target sample of 30 participants | Within 5 months.
  Predetermined count data:
  a. Recruitment to the target sample of 30 participants (15 per arm).
Feasibility - Retention rates | Through participant pathway, on average 18 weeks.
  Progression criteria for retention rates will be evaluated using a 'traffic light system'.
  Green: Retention rate of ≥80%. Retention rates are considered feasible to conduct large scale RCT Amber: Retention rate between 41-79%. Explore methods of increasing retention rates before proceeding to large scale RCT Red: Retention rate ≤40%. Retention rates are not considered feasible to conduct large scale RCT
Feasibility - Outcome measure completion rates | Through participant pathway, on average 18 weeks.
  Green: Completion of ≥80%. Completion rates of outcome measures are considered feasible to conduct large scale RCT Amber: Completion between 41-79%. Explore methods of increasing outcome measure completion rates before proceeding to large scale RCT.
  Red: Completion ≤40%. Completion rates of outcome measures are not considered feasible to conduct large scale RCT
Feasibility - Adherence to group intervention. | Through group intervention, 10 weeks.
  Completion of the group intervention is operationalised as attending 50% or more of the groups.
  Green: Intervention completed by ≥80% of participants. Percentage of participants considered to have completed the group is considered feasible to conduct large scale RCT Amber: Intervention completed by between 41-79% of participants. Explore methods of increasing intervention completion rates before proceeding to large scale RCT Red: Intervention completed by ≤40% of participants. Percentage of participants considered to have completed the group not considered feasible to conduct large scale RCT
Feasibility - Satisfaction Questionnaire | at 18 weeks
  'Neutral' ratings and positive ratings of 'agree' and 'strongly agree' will indicate acceptability of the intervention.
  Satisfaction questionnaire (SQ) adapted for the current research. The brief measure consists of 5 questions that are rated on a 5-point Likert scale, with total score ranging from 5 to 25 where a higher score indicates a higher level of satisfaction. The questionnaire also provides space to enter free text.
Feasibility - Recruitment to the target sample of between 5 and 10 P-BIFS | within 5 months.
  Predetermined count data
Feasibility - P-BIF adherence to intervention protocol | Week 1 of DBT-informed intervention
  Adherent delivery is defined as meeting ≥90% of checklist. P-BIF attendance at supervision will be recorded as an additional measure of treatment adherence.
  Green: ≥90% of all sessions rated as adherent. Attending ≥90% of supervision sessions Amber: Between 80- 89% of all sessions rated as adherent. Attending 80-89% of supervision sessions Red: ≤79% of all sessions rated as adherent. Attending ≤79% of supervision sessions
Feasibility - P-BIF adherence to intervention protocol | Week 2 of DBT-informed intervention
  Adherent delivery is defined as meeting ≥90% of checklist. P-BIF attendance at supervision will be recorded as an additional measure of treatment adherence.
  Green: ≥90% of all sessions rated as adherent. Attending ≥90% of supervision sessions Amber: Between 80- 89% of all sessions rated as adherent. Attending 80-89% of supervision sessions Red: ≤79% of all sessions rated as adherent. Attending ≤79% of supervision sessions
Feasibility - P-BIF adherence to intervention protocol | Week 3 of DBT-informed intervention
  Adherent delivery is defined as meeting ≥90% of checklist. P-BIF attendance at supervision will be recorded as an additional measure of treatment adherence.
  Green: ≥90% of all sessions rated as adherent. Attending ≥90% of supervision sessions Amber: Between 80- 89% of all sessions rated as adherent. Attending 80-89% of supervision sessions Red: ≤79% of all sessions rated as adherent. Attending ≤79% of supervision sessions
Feasibility - P-BIF adherence to intervention protocol | Week 4 of DBT-informed intervention
  Adherent delivery is defined as meeting ≥90% of checklist. P-BIF attendance at supervision will be recorded as an additional measure of treatment adherence.
  Green: ≥90% of all sessions rated as adherent. Attending ≥90% of supervision sessions Amber: Between 80- 89% of all sessions rated as adherent. Attending 80-89% of supervision sessions Red: ≤79% of all sessions rated as adherent. Attending ≤79% of supervision sessions
Feasibility - P-BIF adherence to intervention protocol | Week 5 of DBT-informed intervention
  Adherent delivery is defined as meeting ≥90% of checklist. P-BIF attendance at supervision will be recorded as an additional measure of treatment adherence.
  Green: ≥90% of all sessions rated as adherent. Attending ≥90% of supervision sessions Amber: Between 80- 89% of all sessions rated as adherent. Attending 80-89% of supervision sessions Red: ≤79% of all sessions rated as adherent. Attending ≤79% of supervision sessions
Feasibility - P-BIF adherence to intervention protocol | Week 6 of DBT-informed intervention
  Adherent delivery is defined as meeting ≥90% of checklist. P-BIF attendance at supervision will be recorded as an additional measure of treatment adherence.
  Green: ≥90% of all sessions rated as adherent. Attending ≥90% of supervision sessions Amber: Between 80- 89% of all sessions rated as adherent. Attending 80-89% of supervision sessions Red: ≤79% of all sessions rated as adherent. Attending ≤79% of supervision sessions
Feasibility - P-BIF adherence to intervention protocol | Week 7 of DBT-informed intervention
  Adherent delivery is defined as meeting ≥90% of checklist. P-BIF attendance at supervision will be recorded as an additional measure of treatment adherence.
  Green: ≥90% of all sessions rated as adherent. Attending ≥90% of supervision sessions Amber: Between 80- 89% of all sessions rated as adherent. Attending 80-89% of supervision sessions Red: ≤79% of all sessions rated as adherent. Attending ≤79% of supervision sessions
Feasibility - P-BIF adherence to intervention protocol | Week 8 of DBT-informed intervention
  Adherent delivery is defined as meeting ≥90% of checklist. P-BIF attendance at supervision will be recorded as an additional measure of treatment adherence.
  Green: ≥90% of all sessions rated as adherent. Attending ≥90% of supervision sessions Amber: Between 80- 89% of all sessions rated as adherent. Attending 80-89% of supervision sessions Red: ≤79% of all sessions rated as adherent. Attending ≤79% of supervision sessions
Feasibility - P-BIF adherence to intervention protocol | Week 9 of DBT-informed intervention
  Adherent delivery is defined as meeting ≥90% of checklist. P-BIF attendance at supervision will be recorded as an additional measure of treatment adherence.
  Green: ≥90% of all sessions rated as adherent. Attending ≥90% of supervision sessions Amber: Between 80- 89% of all sessions rated as adherent. Attending 80-89% of supervision sessions Red: ≤79% of all sessions rated as adherent. Attending ≤79% of supervision sessions
Feasibility - P-BIF adherence to intervention protocol | Week 10 of DBT-informed intervention
  Adherent delivery is defined as meeting ≥90% of checklist. P-BIF attendance at supervision will be recorded as an additional measure of treatment adherence.
  Green: ≥90% of all sessions rated as adherent. Attending ≥90% of supervision sessions Amber: Between 80- 89% of all sessions rated as adherent. Attending 80-89% of supervision sessions Red: ≤79% of all sessions rated as adherent. Attending ≤79% of supervision sessions

SECONDARY OUTCOMES:
Change in scores on the Clinical Outcomes of Routine Evaluation -10 | Between week 1 and week 18
  A 10-item measure of psychological distress and a routine psychological therapies recovery outcome measure.
  Scores are presented as a total score (0 to 40) as well as a mean score (between 0 - 4). Higher scores indicate higher levels of general psychological distress, where a total score of 11 or above is within the clinically significant range.
Change in ratings on DIALOG Scale | Between week 1 and week 18
  An 11-item self-report measure of satisfaction across 8 domains providing a score for subjective quality life and treatment satisfaction.
  The mean of the eight items on satisfaction with different life domains forms the subjective quality of life score. The mean of the three items on satisfaction with treatment components forms the treatment satisfaction score. Scores below four reflect explicit dissatisfaction, whereas scores above four reflect explicit satisfaction. Scores of four are the neutral middle point.
Change in scores on Difficulties with Emotional Regulation Scale- 16 | Between week 1 and week 18
  A 16-item measure designed to assess five domains of and overall emotion regulation difficulties.
  Total scores on the DERS-16 can range from 16 to 80, with higher scores reflecting greater levels of emotion dysregulation.
Change in scores on DBT- Ways of Coping Checklist - DBT Skills Subscale | Between week 1 and week 18
  A 38-item self-report measure of DBT skills use. 38 items are rated on a 4-point Likert scale ranging from 0 ( never used ) to 3 ( regularly used ). Higher total scores indicate higher use of of DBT skills use.
Change in score on Distress Tolerance Scale | Between week 1 and week 18
  a 15-item measure assessing the perceived capacity to experience and withstand emotional distress.
  Items are rated on a 5-point Likert scale (5=Strongly disagree to 1=Strongly agree), with higher scores corresponding to greater levels of distress.

CONTACTS AND LOCATIONS:
Locations (1):
- South London and Maudsley NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No